CLINICAL TRIAL: NCT05326087
Title: A Randomized Control Trial to Compare the Euploid Rate of Blastocyst Between the PPOS (Progestin-primed Ovarian Stimulation) Protocol and the Gonadotropin-releasing Hormone (GnRH) Antagonist Protocol in Women With PCOS (Polycystic Ovary Syndrome) Undergoing PGT-A (Preimplantation Genetic Testing for Aneuploidy)
Brief Title: Comparison of the Euploid Rate of Blastocyst Between PPOS and GnRH Antagonist Protocol in Women With PCOS Undergoing PGT-A
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI 2022-03
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Preimplantation Genetic Testing; Progestin-primed Ovarian Stimulation; Polycystic Ovarian Syndrome; GnRH Antagonist
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antagonist group (Active Comparator): Women will receive antagonist (Cetrotide 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Interventions: Drug: GnRH antagonist
- PPOS group (Experimental): Women will receive oral MPA 10mg qd from Day 3 till the day of ovulation trigger.
  Interventions: Drug: MPA

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger
  Other Names: Cetrorelix
  Arms: Antagonist group
Drug: MPA — oral MPA 10mg qd from Day 3 of ovarian stimulation till the day of ovulation trigger.
  Arms: PPOS group

SUMMARY:
This randomized trial aims to compare the euploid rate of blastocysts between PPOS (progestin-primed ovarian stimulation) and GnRH (gonadotrophin releasing hormone) antagonist protocols in patients with PCOS (polycystic ovary syndrome) undergoing PGT-A (preimplantation genetic testing for aneuploidy). Infertile women with PCOS will be recruited for study after explanation and counseling if they fulfill the inclusion criteria and do not have the exclusion criteria. Eligible women will be randomised into one of the two groups:

Antagonist group: Women will receive antagonist once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.

PPOS group: Women will receive oral MPA (medroxyprogesterone acetate)10mg qd from Day 3 till the day of ovulation trigger.

The primary outcome is the euploidy rate of blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Women age between 20 and 37 years.
* Women diagnosed with PCOS according to the modified Rotterdam criteria: oligomenorrhea or amenorrhea, together with the presence of ≥12 antral follicles (≤9 mm) and/or ovarian volume >10 mL on transvaginal ultrasonographic scanning, and/or clinical/ biochemical hyperandrogenism. Other causes of hyperandrogenism and ovulation dysfunction-including tumours, congenital adrenal hyperplasia, hyperprolactinaemia and thyroid dysfunction-were excluded

Exclusion Criteria:

* Presence of a functional ovarian cyst with E2>100 pg/mL
* Endometriosis grade 3 or higher
* Repeated implantation failure (>=4 embryos replaced or >=2 blastocysts replaced without success)
* Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus uni-cornate, bicornate, or duplex); untreated uterine septum, adenomyosis, submucous myoma, or endo-metrial polyp(s)
* Women who are indicated and planned to undergo PGT-SR (Preimplantation genetic testing for structural rearrangement) or PGT-M (Preimplantation genetic testing for monogenic disorder), for example, parental abnormal karyo-type or diagnosed with monogenic disease;
* Recipient of oocyte donation
* Presence of hydrosalpinx which is not surgically treated

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
euploidy rate | 1 month after oocyte retrieval
  euploidy rate of blastocysts

SECONDARY OUTCOMES:
live birth rate | 1 year after embryo transfer
  deliveries ≥22 weeks gestation with heartbeat and breath of the first frozen embryo transfer
cumulative live birth rate | 1 year after embryo transfer
  cumulative live birth within 6 months of randomization
ongoing pregnancy | 12 weeks' gestation
  a viable pregnancy beyond 12 weeks' gestation of the first frozen embryo transfer
number of oocytes retrieved | 1 day after oocyte retrieval
  number of oocytes retrieved
OHSS（ovarian hyperstimulation syndrome） | 1 month after ovarian stimulation
  Moderate or severe ovarian hyperstimulation syndrome.Ovarian hyperstimulation syndrome (OHSS) is diagnosed and classified according to the Royal College of Obstetricians and Gynaecologists guideline.
  Green-top guideline No.5. Ovarian hyperstimulation syndrome. https://www.rcog.org.uk/en/guidelines-research-services/guidelines/gtg5/ (accessed 26 Feb 2016).
birthweight of newborns | 1 year after embryo transfer
  birthweight of newborns

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Principal Investigator — Shanghai JiAi Genetics & IVF Institute, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available when beginning 3 months and ending 5 years following article publication.
Access Criteria: To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with. Proposals should be sent to lihe198900@163.com.

REFERENCES:
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Lee E, Illingworth P, Wilton L, Chambers GM. The clinical effectiveness of preimplantation genetic diagnosis for aneuploidy in all 24 chromosomes (PGD-A): systematic review. Hum Reprod. 2015 Feb;30(2):473-83. doi: 10.1093/humrep/deu303. Epub 2014 Nov 28. PMID 25432917
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Ehrmann DA, Liljenquist DR, Kasza K, Azziz R, Legro RS, Ghazzi MN; PCOS/Troglitazone Study Group. Prevalence and predictors of the metabolic syndrome in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Jan;91(1):48-53. doi: 10.1210/jc.2005-1329. Epub 2005 Oct 25. PMID 16249284